CLINICAL TRIAL: NCT02111044
Title: A Randomized, Multicenter, Phase II Study to Investigate Efficacy and Safety of ITF2984 in Acromegalic Patients
Brief Title: Phase II Study With ITF2984 in Acromegalic Patients
Acronym: POC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DSC/13/2984/05
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Acromegaly
Keywords: de novo or partial responder to somatostatin analogues
MeSH Terms: conditions — Acromegaly | interventions — Octreotide; Somatostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Octreotide (Active Comparator): Octreotide 100 mcg sc three times daily (t.i.d) for 4 weeks
  Interventions: Drug: Octreotide
- ITF2984 500 mcg (Experimental): ITF2984 500 mcg sc twice a day (b.i.d) for 4 weeks
  Interventions: Drug: ITF2984 500 mcg
- ITF2984 1000 mcg (Experimental): ITF2984 1000 mcg sc b.i.d for 4 weeks
  Interventions: Drug: ITF2984 1000 mcg
- ITF2984 2000 mcg (Experimental): ITF2984 2000 mcg sc b.i.d for 4 weeks
  Interventions: Drug: ITF2984 2000 mcg

INTERVENTIONS:
Drug: Octreotide — octreotide 100 mcg sc t.i.d. for 4 weeks
  Other Names: somatostatin analog
  Arms: Octreotide
Drug: ITF2984 500 mcg — ITF2984 500 mcg sc b.i.d for 4 weeks
  Other Names: somatostatin analog
  Arms: ITF2984 500 mcg
Drug: ITF2984 1000 mcg — ITF2984 1000 mcg sc b.i.d for 4 weeks
  Other Names: somatostatin analog
  Arms: ITF2984 1000 mcg
Drug: ITF2984 2000 mcg — ITF2984 2000 mcg sc b.i.d for 4 weeks
  Other Names: somatostatin analog
  Arms: ITF2984 2000 mcg

SUMMARY:
The purpose of this study is to investigate in acromegalic patients the effect of different doses of ITF2984 on GH and IGF-1 concentrations and to investigate safety and tolerability of three different doses of ITF2984.

DETAILED DESCRIPTION:
The study will enroll patients with active acromegaly, de novo or partial responder to previous treatment with somatostatin analogues. For patients who had previously received medical therapy for acromegaly a washout periods before study entry of 3 months for long-acting formulation of somatostatin analogs, 2 weeks for octreotide sc, 2 months for pegvisomant and/or cabergoline must be foreseen.

Each patient will be randomized and wll remain in the study for about 6 months, and they will attend a visit every two weeks.

The patients will be treated for 4 months in a total, in particular every month of treatment will be followed by a washout period of 2 weeks.

At each month of treatment the patients will receive one of the four treatment as reported below:

Octreotide 100 mcg sc three times daily (t.i.d) for 4 weeks, ITF2984 500 mcg sc twice a day (b.i.d) for 4 weeks, ITF2984 1000 mcg sc b.i.d for 4 weeks, ITF2984 2000 mcg sc b.i.d for 4 weeks. Patients will be randomized using a 4 way crossover design to receive ITF2984 or octreotide at each treatment month. Each patient will receive all of the four treatments overseen in this study.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Patients with active acromegaly due to a pituitary adenoma. Active acromegaly should be confirmed by 2h five point mean GH level higher than 5 mcg/liter, lack of suppression of GH nadir to less than 1 mcg/liter after oral glucose tolerance test, and elevated IGF-1 for age and sex-matched controls.
* Patients aged between 18 to 80 years old inclusive.
* Patients treated with previous surgery and/or medical therapy or previously untreated (de novo). For patients who had previously received medical therapy for acromegaly a washout periods before study entry of 3 months for long-acting formulation of somatostatin analogs and 2 weeks for octreotide sc must be foreseen. Partial responder means a significant decrease (>50%), without achievement of control of GH and/or IGF-1 levels and/or >20 % tumor shrinkage after at least 6 months of SRL therapy.
* Patients with GH level and IGF-1 level for age and sex-matched controls out of range at baseline (GH at baseline > 2.5mcg/l).

Exclusion Criteria:

* Patients undergone pituitary surgery within the prior 6 months.
* Patients who have received pituitary radiotherapy (within last 10 years).
* Patients with additional active malignant disease within the last five years (with the exception of basal cell carcinoma or carcinoma in situ of the cervix)
* Patients with compression of the optic chiasm causing any visual field defect.
* Patients who require a surgical intervention for relief of any sign or symptom associated with tumor compression.
* Patients with uncontrolled diabetes defined as having a fasting glucose > 150 mg/dL (8.3 mmol/L) or HbA1c ≥ 8% (Patients can be rescreened after diabetes is brought under adequate control).
* Patients who have had a significant cardiovascular disease in the three months prior to inclusion such as congestive heart failure (NYHA [New York Heart Association] class III or IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation, sustained clinically significant bradycardia, advanced heart block, or with a history of acute myocardial infarction.
* A marked baseline prolongation of QT/QTc interval i.e. a mean QT/QTc >450ms after 3 consecutive measurements at least 5 minutes apart.
* Patients with abnormal coaugulation, Prothrombin time (PT), activated partial thromboplastin time (PTT) elevated by 30% above normal limits.
* Symptomatic cholelithiasis, gallstone or chronic liver disease.
* Patients who have a history or presence at the moment of the screening visit of pancreatitis.
* Clinically significant GI, renal or hepatic disease (in the opinion of investigator).
* AST and/or ALT>2ULN.
* Severely reduced renal function (serum creatinine >2.0 mg/dl or 176µmol/L)
* Active HBV and/or active HCV infection.
* Patients who have a history of alcohol or drug abuse in the six-month period prior to the enrollment visit.
* Known hypothyroidism or hypocortisolism not adequately treated with a stable dose of thyroid or steroid hormone replacement therapy for at least the previous 3 months.
* Known hypersensitivity to any of the study medications, or components thereof or a history of drug or other allergy that in the opinion of the Investigator contraindicates their participation.
* Female patients who are pregnant or lactating, and female patient who are of childbearing potential or male patient with female partners of childbearing potential who do not accept the contraception requirements reported in the protocol.
* Patients who have participated in any clinical investigation with an Investigational drug within 3 months before study entry.
* Current or recent (< 2 months) therapy with pegvisomant or cabergoline.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
effect of treatment on GH and IGF-1 | 4 weeks
  To investigate the effect of treatment on GH and IGF-1 concentrations

SECONDARY OUTCOMES:
reduction in (random) GH < 1.0 mcg/l and/or normalization of IGF-1 | 4 weeks
  To investigate the biochemical response, defined as a reduction in (random) GH < 1.0 mcg/l and/or normalization of IGF-1.
reduction of GH to no more than 2.5 mcg/l and/or normalization of IGF-1 | 4 weeks
  To investigate the biochemical response, defined as a reduction of GH to no more than 2.5 mcg/l and/or normalization of IGF-1.
signs and symptoms of acromegaly | 4 weeks
  To evaluate variation of signs and symptoms of acromegaly at the end of each month of treatment in comparison with basal status.
PK profile of ITF2984 and Octreotide | 4 weeks
  To investigate the pharmacokinetic (PK) profile of ITF2984 and Octreotide
dose-response effect of ITF2984 on GH and IGF1 circulating levels | 4 weeks
  To compare the effects on GH and IGF1 circulating levels of different doses of ITF2984
effects of ITF2984 vs Octreotide on GH and IGF1 circulating levels | 4 weeks
  To compare the effects on GH and IGF1 circulating levels of ITF2984 and Octreotide

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bettica, MD, Study Director — Italfarmaco
Locations (26):
- Czechia (2):
  - St. Anne University Hospital, Brno
  - University Hospital Hradec Kralove, Hradec Králové
- France (2):
  - Université Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital de la TIMONE, Marseille
- Hungary (4):
  - Az MH Honvédkórház, Budapest
  - Semmelweis University, Budapest
  - University of Pecs, Pécs
  - University of Szeged, Szeged
- Italy (7):
  - Presidio Ospedaliero di Montichiari, Brescia
  - Policlinico G. Martino, Messina
  - Fondazione Policlinico IRCCS, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Università Federico II, Napoli
  - Università di Pisa, Pisa
  - San Giovanni Battista Molinette, Torino
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Erasmus Medisch Centrum, Rotterdam
- Poland (3):
  - University Children's Hospital of Cracow, Krakow
  - Klinika Endokrynologii Centrum Medycznego Kształcenia Podyplomowego, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny, Wroclaw
- Romania (3):
  - Institutul de Endocrinologie C.I.Parhon, Sectia clinica de endocrinologie II, Bucharest
  - Institutul de Endocrinologie C.I.Parhon, Sectia clinica de endocrinologie I, Bucharest
  - Institutul de Endocrinologie C.I.Parhon, Sectia clinica de endocrinologie VI, Bucharest
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - Clinical center of Nis, Niš
- Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, Spain